CLINICAL TRIAL: NCT05421611
Title: A Phase III, Multicenter, Double Blind, Randomized Study of SII Yellow Fever Vaccine to Compare Safety and Immunogenicity With STAMARIL
Brief Title: A Study of SII Yellow Fever Vaccine to Compare Safety and Immunogenicity With STAMARIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: YWF:03
Record Dates: First submitted 2022-06-13; First posted 2022-06-16 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Yellow Fever
MeSH Terms: conditions — Yellow Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SII-YFV (Experimental): Live attenuated Yellow Fever Virus (17D-213 Strain) not less than 1000 IU/dose propagated in specific pathogen-free chick embryos
  Diluent: 0.5 mL of sterile water for injection
  Interventions: Biological: SII-YFV
- STAMARIL (Active Comparator): Live attenuated Yellow Fever Virus (17D-204 Strain) not less than 1000 IU/dose produced in specified pathogen-free chick embryos
  Solvent: Sodium Chloride 2.0 mg; Water for injections up to 0.5 mL
  Interventions: Biological: STAMARIL

INTERVENTIONS:
Biological: STAMARIL — STAMARIL® contains the 17D-204 vaccine strain, which is used in many currently produced yellow fever vaccines. STAMARIL is specific pathogen free embryonated hen's egg based and is prepared by harvesting and stabilizing the virus collected from the homogenized chicken embryos infected with YF vaccine virus.
  STAMARIL® will be used as a comparator in the study. It is a live, attenuated, freeze-dried (lyophilized) vaccine and is to be reconstituted with solvent.
  Arms: STAMARIL
Biological: SII-YFV — SII-YFV contains the 17D-213 vaccine strain, a derivative of 17D-204 strain which is used in many currently produced yellow fever vaccines. SIIPL imported the YF WHO Primary Seed Virus lot 213-77 from National Institute for Biological Standards and Control (NIBSC) for preparation of the master seed virus, working seed virus and the vaccine. The SII-YFV is specific pathogen free embryonated hen's egg based and is prepared by harvesting and stabilizing the virus collected from the homogenized chicken embryos infected with YF working seed virus.
  SII-YFV will be provided in vial presentation for the study. It is a live, attenuated, freeze-dried (lyophilized) vaccine and is to be reconstituted with sterile water for injection.
  Arms: SII-YFV

SUMMARY:
The study is designed as a Phase III, double-blind, multicenter, randomized, active-controlled, parallel-group design in which two groups of participants will receive either SII-YFV or STAMARIL® - a licensed and WHO pre-qualified YFV. The study will start only after the approval from the applicable ethics committees and national regulatory agencies.

DETAILED DESCRIPTION:
There will be three scheduled visits during the study. A screening and vaccination visit (Day 0) followed by additional study visits on Day 28 and on Day 180 post-vaccination. Throughout the study, participants/parent/guardian will be encouraged to contact the study team if the participant is unwell and the study team will additionally maintain contact with study participants. The participant or parent/guardian will be contacted telephonically on Day 90 to enquire about participant's health and occurrence of any serious adverse events (SAEs). Active surveillance for vaccine reactogenicity will be conducted in reactogenicity cohort from the time of vaccination (Day 0) until Day 10 following vaccination. Unsolicited AE will be collected from all study participants until Day 28 post vaccination. SAEs will be collected from all participants throughout the study (to Day 180).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged ≥ 1 year
2. Healthy volunteers as determined by medical history and clinical examination
3. Participants willing to adhere to the protocol requirements and to provide informed consent for participants ≥ 18 years of age. For participants < 18 years of age, parental/guardian ability and willingness to provide informed consent (as per local requirements/procedures) and additional informed assent from participants, as appropriate for participating community (i.e. participants at least 7 years of age in Kenya)
4. Intend to remain residing in study area throughout the study participation
5. Female participants of childbearing potential* must have practiced adequate contraception** and agree to continue adequate contraception till Day 28 post-vaccination.
6. Female participants of childbearing potential must have a negative pregnancy test within 24 hours prior to IP administration.
7. Be willing to avoid the use of traditional/herbal local medications and treatments for the duration of the study

Exclusion Criteria:

1. Fever (> 37.5°C) or any clinically significant acute infection at time of vaccination [Temporary exclusion criteria - participants may be re-screened at least 48 hours after the last recorded fever]
2. Use of systemic (oral or parenteral) antibiotics or antiviral agents within the past 7 days. [Temporary exclusion criteria - participants may be re-screened at least 7 days after last dose of antibiotics or antiviral agents]
3. Use of traditional/herbal local medications and treatments in the past 7 days [Temporary exclusion criteria - participants may be re-screened at least 7 days after last consumption of traditional/herbal local medications and treatment]
4. Previous history of laboratory confirmed infection with yellow fever and other flaviviruses e.g., dengue fever, tick-borne-encephalitis (TBE), Japanese encephalitis (JE), West Nile virus (WNV), zika virus, etc.
5. Previous vaccination against yellow fever, TBE, JE, or dengue fever.
6. Receipt of any vaccine within past 28 days or planned vaccination until completion of Day 28 visit
7. Known or suspected impairment of immunological function based on medical history and physical examination.
8. Presence of any systemic disorder (cardiovascular, pulmonary, hepatic, renal, gastrointestinal, hematological, endocrine, immunological, dermatological, neurological, cancer, or autoimmune disease) as determined by medical history and / or physical examination which would compromise the participant's health or is likely to result in nonconformance to the protocol
9. History of chronic administration (defined as more than 14 consecutive days) of immunosuppressant (> 0.5 mg/kg/day of prednisolone or equivalent) or other immune modifying drugs including the use of glucocorticoids. The use of topical/inhaled/per nasal glucocorticoids will be permitted.
10. A known hypersensitivity to any of the vaccine components (including gelatin, eggs, egg products, or chicken protein) or history of a life-threatening reaction to any past vaccine.
11. Receipt of any immunoglobulin therapy and / or blood products in the past 60 days or planned administration until completion of Day 28 visit.
12. Participation in a drug research study, involving investigational products, within past 3 months or planned participation during the entire study period
13. Receipt of any investigational or unlicensed medication (drug or vaccine) in the preceding 28 days, or planned use until completion of Day 28 visit
14. Uncontrolled coagulopathy or blood disorder contraindicating subcutaneous injections or blood sampling
15. Be an employee of, or direct descendant (child or grandchild) of any person employed by the investigator or sponsor.
16. Pregnant or lactating women
17. Requirement of Yellow Fever vaccination certificate for travelling purpose
18. History of thymus dysfunction including myasthenia gravis, thymoma, thymectomy
19. History or presence of significant alcoholism or drug abuse in the past one year
20. Major congenital or genetic defect
21. Any other condition which in the opinion of the investigator will jeopardize the safety of the participant or compromise the assessment of the study objectives

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1824 (Actual)
Dates: Start 2023-05-11 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
YF neutralizing antibody (NAb) seroconversion rates | 28 days post vaccination
  NI comparison for primary objective of the study will be based on seroconversion rate at 28 days post vaccination i.e. percentage of participants achieving seroconversion. Seroconversion is defined as a fourfold increase in neutralizing antibody from baseline.

SECONDARY OUTCOMES:
GMTs achieved with SII-YFV versus STAMARIL | 28 days post vaccination
  To compare the YF NAb geometric mean titres (GMTs) generated following SII-YFV to those generated following STAMARIL®.

CONTACTS AND LOCATIONS:
Locations (2):
- Kenya (2):
  - Victoria Biomedical Research Institute (VIBRI) - Kisumu County Referral Hospital, Kisumu
  - Kenya Medical Research Institute/ Centre for Research Disease Research (CRDR), Nairobi

IPD SHARING:
Plan to Share IPD: Yes
Data collected from this study will be made available upon publication to members of the scientific and medical community for non-commercial use only, upon email request to the corresponding author. other study details are available on clinicaltrials.gov.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 6 months of publication of the study data
Access Criteria: Local regulatory authorities, ethics committee